CLINICAL TRIAL: NCT00999622
Title: CD4 Count And Risk Of Infection In Patients With Brain Tumors
Brief Title: Study of Blood Samples and Risk of Infection in Patients With Newly Diagnosed Malignant Supratentorial Astrocytoma
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH); North American Brain Tumor Consortium (Other)
Responsible Party: Sponsor
Other Study IDs: NABTT-0305 CDR0000363636; U01CA062475 (NIH); NABTT-0305
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Brain and Central Nervous System Tumors; Infection
Keywords: infection; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult giant cell glioblastoma; adult gliosarcoma; adult oligodendroglioma; adult glioblastoma; adult diffuse astrocytoma; adult pilocytic astrocytoma; adult pineal gland astrocytoma; adult subependymal giant cell astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Infections; Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Other: laboratory biomarker analysis
Other: questionnaire administration

SUMMARY:
RATIONALE: Gathering information over time from laboratory tests of patients with newly diagnosed malignant supratentorial astrocytoma may help doctors learn more about the effect of treatment on white blood cell count and the risk of infection.

PURPOSE: This clinical trial is studying blood samples and risk of infection in patients with newly diagnosed malignant supratentorial astrocytoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the frequency and severity of decreases in CD4 counts as a function of therapy in patients with newly diagnosed malignant astrocytoma.
* Determine whether the decrease in CD4 counts is a significant predictor of infections or adverse outcomes in these patients.

OUTLINE: This is a multicenter study.

Patients undergo monthly collection of blood for serial CD4 counts and heme-8 with differential for 1 year for quantitative analysis. Patients also complete a monthly questionnaire about infections and antibiotic use.

Patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 125 patients (100 with high-grade disease and 25 with low-grade disease) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary malignant brain tumor in 1 of the following groups:

  * High grade (grade III or IV) supratentorial glioma receiving antineoplastic treatment and with 1 of the following histologies:

    * Anaplastic astrocytoma
    * Glioblastoma multiforme (giant cell glioblastoma or gliosarcoma)
    * Anaplastic oligodendroma
  * Low grade (grade I or II) supratentorial glioma not planning to receive treatment of any kind (including steroids) and with 1 of the following histologies:

    * Astrocytoma
    * Oligodendroglioma

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* No HIV positivity

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for brain tumor except polifeprosan 20 with carmustine implant (Gliadel® wafer)
* No prior cranial radiotherapy or radiotherapy for brain tumor
* No prior immunotherapy or biologic agents for brain tumor, including any of the following:

  * Immunotoxins
  * Immunoconjugates
  * Peptide receptor antagonists
  * Interleukins
  * Interferons
  * Tumor-infiltrating lymphocytes
  * Lymphokine-activated killer cell therapy
  * Gene therapy
  * Antisense therapy
* No prior hormonal therapy for brain tumor

  * More than 14 days since prior and no concurrent steroid therapy for patients with low-grade (grade I or II) astrocytoma
  * Prior glucocorticoid therapy allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High grade and low grade
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2004-07; Primary Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of decreases in CD4 counts | 1 year
Determination of decrease in CD4 counts as significant predictor of infections or adverse outcomes | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A. Grossman, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins